CLINICAL TRIAL: NCT00099255
Title: A Phase II Multi-Dose Study of SGN-30 (Anti-CD30 mAb) in Patients With Primary Cutaneous Anaplastic Large Cell Lymphoma, Large Cell Transformation of Mycosis Fungoides, and Lymphomatoid Papulosis
Brief Title: Study of SGN-30 (Anti-CD30 mAb) in Patients With Primary Cutaneous Anaplastic Large Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SG030-0004; NCT00118079 (obsolete NCT alias)
Record Dates: First submitted 2004-12-10; First posted 2004-12-10 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Large Cell Lymphoma
Keywords: Keyword?; Primary Cutaneous Anaplastic Large Cell Lymphoma; Large Cell Transformation of Mycosis Fungoides; Lymphomatoid Papulosis
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Primary Cutaneous Anaplastic Large Cell; Lymphomatoid Papulosis | interventions — Brentuximab Vedotin

INTERVENTIONS:
Drug: SGN-30

SUMMARY:
This multi-center, phase II study will be conducted to define the toxicity profile and antitumor activity of SGN-30 in patients with pcALCL and other closely related lymphoproliferative disorders.

ELIGIBILITY:
Inclusion Criteria

* Patients must have a definite diagnosis.
* Patients must be histologically confirmed CD30 positive within 3 months of enrollment
* Patients with pcALCL must have target lesions present for at least 1 month without spontaneous regression
* pcALCL patients must have failed treatment with local radiation therapy, or failed systemic therapy of a single agent
* Patients must be considered an eligible candidate for systemic therapy as determined by the investigator
* All patients must have a three week wash-out from previous treatments, unless in the opinion of the investigator it is not in the best interest of the patient, at which point the individual case must be discussed with the medical monitor prior to enrollment.
* Patients must have an ECOG performance status of < 2 (Appendix B) and a life expectancy > six months.
* Patients must be at least 18 years of age.
* Patients must be available for periodic blood sampling, study-related assessments, and management of toxicity at the treating institution.
* Females of childbearing potential must have a negative HCG pregnancy test result within three days of enrollment. All patients must agree to use an effective contraceptive method during the course of the study.
* Patients must give written informed consent.
* Required baseline laboratory data: Absolute neutrophil count greater than or equal to to 1,000/mm3, Platelet count greater than or equal to 75,000/mm3, Serum bilirubin less than or equal to 1.5 times ULN, Serum creatinine less than or equal to 1.5 times ULN, BUN less than or equal to 1.5 times ULN, SGOT less than or equal to 2.5 ULN, SGPT less than or equal to 2.5 ULN

Criteria for Exclusion

* Patients with Sezary syndrome, or any type of lymphoproliferative disease other than pcALCL, T-MF or LyP
* Patients with systemic ALCL or extracutaneous involvement of cutaneous ALCL
* Patients with known active systemic viral, bacterial, or fungal infection
* Patients who are known to be HIV, Hepatitis B, or Hepatitis C positive
* Patients who have been treated previously with any anti-CD30 antibody
* Patients with a known hypersensitivity to recombinant proteins or any excipient contained in the drug formulation
* Patients with a history of other malignancies during the past five years with the exception of adequately treated basal or squamous cell skin cancer or cervical carcinoma in situ
* Patients with symptomatic cardiac disease including ventricular dysfunction, coronary artery disease, or arrhythmias
* Patients who are pregnant or breastfeeding
* Patients with any serious underlying medical condition that would impair their ability to receive or tolerate the planned treatment
* Patients with dementia or altered mental status that would preclude understanding and rendering of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-09; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
To determine the objective response rate in patients with pcALCL, T-MF, and LyP
To determine the duration of response in patients treated with SGN-30
To investigate the toxicity profile of SGN-30

SECONDARY OUTCOMES:
To provide preliminary estimates of disease-free and overall survival rates in pcALCL and T-MF patients treated with SGN-30
To determine the immunogenicity of SGN-30

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California at Los Angeles, Los Angeles, California
  - Stanford University, Stanford, California
  - Yale, New Haven, Connecticut
  - Northwestern Universtiy, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Johns Hopkins, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Memorial Sloan-Kettering, New York, New York
  - Cleveland University, Cleveland, Ohio
  - Kaiser Permanente - Oncology Research, Portland, Oregon
  - Vanderbilt University, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Duvic M, Reddy SA, Pinter-Brown L, Korman NJ, Zic J, Kennedy DA, Lorenz J, Sievers EL, Kim YH. A phase II study of SGN-30 in cutaneous anaplastic large cell lymphoma and related lymphoproliferative disorders. Clin Cancer Res. 2009 Oct 1;15(19):6217-24. doi: 10.1158/1078-0432.CCR-09-0162. Epub 2009 Sep 29. PMID 19789316
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/19789316